CLINICAL TRIAL: NCT03552458
Title: Effects of Probiotics Intake on Oral Microbiome and Mucosa Inflammation in Patients With Cytotoxic Therapy Induced Oral Mucositis: A Pilot Study
Brief Title: Effects of Probiotics in Preventing Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017/00508
Record Dates: First submitted 2018-04-15; First posted 2018-06-11 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Head-and-neck Cancer
Keywords: oral mucositis; probiotics; anti-neoplastic chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Intervention Model Description: randomized double blind prospective placebo controlled clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LR group (Experimental): Lactobacillus Reuteri Oral Solution [BioGaia]
  Interventions: Drug: Lactobacillus Reuteri Oral Solution [BioGaia]
- Placebo group (Placebo Comparator): Placebos: The control agent will not contain the active agent
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lactobacillus Reuteri Oral Solution [BioGaia] — BioGaia Lactobacillus Reuteri drops
  Other Names: Biogaia Prodentis
  Arms: LR group
Drug: Placebos — Placebo will be identical in physical appearance and color to the study agent and will be made by the manufacturer
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
The study will be a randomized double blind prospective placebo controlled clinical study and aims to determine the therapeutic efficacy of Probiotics in Oral Mucositis pathogenesis in patients undergoing head and neck radiotherapy.

DETAILED DESCRIPTION:
The study will be a randomized double blind prospective placebo controlled clinical study (Clinical Trial phase II) of 50 patients (25 in LR group, 25 in placebo group) with a confirmed cancer diagnosis requiring head and neck radiotherapy with a minimum dose of 6000cGy.

Patients will be randomly assigned to either of the treatment arms in a 1:1 ratio. The active agent; Lactobacillus reuteri Prodentis (Biogaia ®) will be supplied in droplet form by Pharma forte Singapore Pte Ltd and dosage used will be as recommended by manufacturer (5 drops/time twice a day which is equivalent to 4 X 108 CFU of live bacteria). The control agent will be identical in physical appearance and color to the study agent and will be made by the manufacturer.

Patients assigned to either LR group or placebo group will start from the first day of radiotherapy and continued until 2-week post radiation (approximately 8-9 weeks). Patients will be instructed to use the LR droplets twice a day according to manufacturer's instructions; once in the morning after breakfast and the other just before bedtime and to avoid any food/drinks 30 minutes before and after usage. Compliance with treatment will be elicited and recorded.

The dose selection is based on manufacturer's recommendations and is safe for use during pregnancy and breastfeeding. However, this is not an issue in this population as none of the patients should be pregnant or breastfeeding while receiving radiation and anti-neoplastic chemotherapy.

The PI will serve as the auditor for data quality assurance on a quarterly basis.Data collected on paper will be stored in the principal investigator's locked cabinet. Data will be entered into Microsoft Excel™ (2007) and double entered for accuracy. Data will be kept in a password secured portable computer and backed up to dedicated local back-up drive every week. Only group statistics will be reported. The database will only be accessible to investigators involved in and approved for the study. All data will be kept for 6 years after study completion to access data for publication of the work done, after which data will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are 21 years of age or older
2. histological diagnosis of head and neck carcinoma available
3. undergoing head and neck radiotherapy of at least 6000cGY
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
5. no known allergy to Biogaia
6. able to give written informed consent, or have written consent given on their behalf.

Exclusion Criteria:

1. patients who cannot use the products or have it administered to them
2. patients with existing conditions predisposing to oral ulcer formation
3. patients with mucositis at baseline (prior to initiation of treatment)
4. previous radiotherapy to the head and neck region
5. female patients who are pregnant or breastfeeding
6. patients who have central venous catheters
7. patients who have impaired intestinal epithelial barrier
8. patients who have cardiac valvular disease
9. unable to give written informed consent, or are unable to have written consent given on their behalf.
10. inability to converse in English or Mandarin
11. severe immunosuppression (Absolute Neutrophil Count of less than 1500 cells/µL)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis (OM) Severity Assessment | Weekly review from baseline (Day 1 of Radiation) to 14 days after last radiation treatment
  To assess the severity of OM using Oral Mucositis Assessment Scale (OMAS)
Oral Mucositis (OM) Severity Assessment | Weekly review from baseline (Day 1 of Radiation) to 14 days after last radiation treatment
  To assess the severity of OM (Grade 0-4) using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0
Duration of Oral Mucositis (OM) | Weekly review from baseline (Day 1 of Radiation) to 14 days after last radiation treatment
  To assess the number of days of OM experienced i.e. start of OM still resolution of OMM
Pain Severity of OM | Weekly review from baseline (Day 1 of Radiation) to 14 days after last radiation treatment
  Visual Analogue Scale (0-10)
Quality of Life post Radiation | Daily Patient Completed Questionnaire from baseline (Day 1 of Radiation) to 14 days after last radiation treatment
  Composite score using the Oral Mucositis Daily Questionnaire (8 Item questionnaire)

SECONDARY OUTCOMES:
Oral Bacteria Analysis and Gene Expression Analysis | Change between baseline and Week 4
  Oral samples will be collected at 2 time points: baseline (before start of head and neck radiotherapy) and at week 4 (Visit 5, midpoint) of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hong, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goh CE, Williams R, Gupta N, Ho F, Islam I, Lai CWM, Tan KS, Hong CHL. Effect of Limosilactobacillus reuteri Probiotic on Oral Mucositis in Patients Undergoing Head and Neck Radiation: A Randomised Trial. Oral Dis. 2025 Aug 31. doi: 10.1111/odi.70083. Online ahead of print. PMID 40887814